CLINICAL TRIAL: NCT01939405
Title: Use of the Built Environment to Promote Physical Activity in Children.
Brief Title: Children's Use of the Built Environment for Physical Activity
Acronym: CUBES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nicolas M. Oreskovic, MD, MPH, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2010P001480; K23HL103841 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight; Physical Activity; Built Environment; counseling
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard physical activity counseling (No Intervention)
- built environment use counseling (Experimental): personalized counseling on active use of the built environment
  Interventions: Behavioral: built environment use counseling

INTERVENTIONS:
Behavioral: built environment use counseling
  Arms: built environment use counseling

SUMMARY:
The study aims are to develop and test the feasibility of a pediatric physical activity intervention that incorporates personal information on use of the built environment, and test the intervention's preliminary efficacy at increasing physical activity. The investigators hypothesize that it will be feasible to incorporate and measure changes in empiric GIS (geographic information system), GPS (global positioning system), and accelerometer feedback in the office setting as demonstrated by: i) Completeness of GPS and accelerometer data collection (primary measure of feasibility), ii) Participation rates among adolescents in the intervention group compared to the control group, and iii) Acceptability to patients as measured by adolescent satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 10-16 years
* BMI > 85th percentile for age and sex

Exclusion Criteria:

* Physical conditions impairing ambulation
* Adolescents who do not speak English
* Adolescents who have missed more than 2 scheduled doctor's appointments during the past 5 years
* Adolescents who are receiving any other form of physical activity counseling/intervention at the time of enrollment

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Oreskovic, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Revere HealthCare Center, Revere, Massachusetts, United States

REFERENCES:
- [Derived] Oreskovic NM, Winickoff JP, Perrin JM, Robinson AI, Goodman E. A Multimodal Counseling-Based Adolescent Physical Activity Intervention. J Adolesc Health. 2016 Sep;59(3):332-337. doi: 10.1016/j.jadohealth.2016.03.012. Epub 2016 May 24. PMID 27235377

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Physical Activity Counseling: standard pedatric physical activity counseling
- Built Environment Use Counseling: personalized counseling on active use of the built environment
  built environment use counseling
Period: Overall Study
Arm/Group | Standard Physical Activity Counseling | Built Environment Use Counseling
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard Physical Activity Counseling: standard pediatric physical activity counseling
- Total: Total of all reporting groups
Arm/Group | Standard Physical Activity Counseling | Built Environment Use Counseling | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (1.0) | 12.2 (1.6) | 11.9 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 15 | 13 | 28
  Race/Ethnicity: Black | 3 | 1 | 4
  Race/Ethnicity: Hispanic | 8 | 10 | 18
  Race/Ethnicity: Asian | 2 | 1 | 3
  Race/Ethnicity: Multi/Other | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
BMI percentile [Mean (Standard Deviation); unit: BMI percentile] | 94 (3.9) | 94 (3.9) | 94 (3.9)
parental education [Count of Participants; unit: Participants]
  High School or less | 9 | 11 | 20
  Associates degree or College | 16 | 18 | 34
  Graduate Education | 4 | 1 | 5
  missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Moderate to Vigorous Physical Activity (MVPA)
Description: Short-term change in MVPA from baseline to post-intervention
Time Frame: Immediately post-intervention
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Physical Activity Counseling | Built Environment Use Counseling
Number analyzed (Participants) | 27 | 28
minutes | -1.9 [-14.1 to 3.7] | 1.07 [-14.7 to 21.4]

2. Secondary Outcome: Moderate-to-Vigorous Physical Activity (MVPA)
Description: Longer term change in MVPA from baseline to 3-4 months post intervention
Time Frame: 4 months from baseline
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Physical Activity Counseling | Built Environment Use Counseling
Number analyzed (Participants) | 27 | 28
minutes | 0.5 [-22.7 to 4.1] | 6.3 [-31.1 to 11.8]

3. Secondary Outcome: Sedentary Time
Description: Short-term change in sedentary (non-active) time from baseline to post-intervention, objectively measured using accelerometers
Time Frame: Immediately post-intervention
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | Standard Physical Activity Counseling | Built Environment Use Counseling
Number analyzed (Participants) | 27 | 28
minutes | 11.1 (73.9) | 5.8 (86.3)

4. Secondary Outcome: Sedentary Time
Description: Longer-term change in sedentary (non-active) time from baseline to 3-4 months post-intervention, objectively measured using accelerometers.
Time Frame: 4 months from baseline
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | Standard Physical Activity Counseling | Built Environment Use Counseling
Number analyzed (Participants) | 27 | 28
minutes | -22.9 (75.6) | -4.4 (91.3)

ADVERSE EVENTS:
Description: The meaning of "0" Total Number of Participants at Risk (e.g., "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events) were not monitored/assessed.
Arm/Group | Standard Physical Activity Counseling | Built Environment Use Counseling
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small sample size, single office setting, short term (4 months) follow-up, multi-component intervention including financial incentives and text messages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No